CLINICAL TRIAL: NCT06248385
Title: The Correlation of the Lower Placental Edge Thickness in Relation to Gestational Age at Delivery by Using Ultrasonography in Patients With Placenta Previa Accreta; A Prospective Cohort Study
Brief Title: Lower Placental Edge Thickness in Relation to Gestational Age at Delivery in Placenta Accreta (Prospective Cohort Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: TVS in placenta accreta
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-01

CONDITIONS: Placenta Accreta
Keywords: Placental edge thickness; Placenta Accreta; Preterm delivery
MeSH Terms: conditions — Placenta Accreta; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 2D ultrasound — 2D TVUS

SUMMARY:
The aim of our study is to determine correlation between lower placental edge thickness measured by ultrasound and gestational age at delivery and predict the risk of emergency preterm birth in patients having placenta previa accreta.

DETAILED DESCRIPTION:
In pregnant women with placenta previa accreta, the lower placental edge thickness measured by ultrasound may correlate with gestational age at delivery and predict emergency preterm cesarean delivery. Thick lower placental edge is thought to be responsible for emergency preterm birth.

All women who meet the inclusion criteria will undergo full assessment to identify eligible women.

This assessment will include:

Detailed History:Personal history: age, duration of marriage, smoking. Present history: any current medical or surgical diseases and current medication.

Past medical history: history of medical disorders like diabetes and hypertension.

Surgical history: previous uterine surgery and previous cesarean section. Menstrual history: Regularity, duration, amount, LMP. Contraceptive history: Previous used methods, any complications from any used method.

Obstetric history: Gravidity, parity, abortions, living, mode of delivery, date of the last delivery, gestational age and any obstetric complications.

Clinical examination:

General examination:

Assessment of patient general condition. vital data (pulse, blood pressure, temperature). Color of complexion e.g.: pallor in anemic patients.

Abdominal examination:

Inspection: globular abdomen, previous scar. Palpation: abdominal pain, tenderness, rigidity, uterine consistency, symphysio-fundal height (SFH) measurement, fetal lie, fetal presentation.

Auscultation: fetal heart sounds. Pelvic examination:Will not be done.

Ultrasound examination:

2D ultrasound will be carried out trans-abdominally to assess fetal viability and number, placental location, determine gestational age and fetal anomalies and calculate exact amniotic fluid index (AFI).

TVUS and placental bed Doppler will be done to confirm exact placental site and confirm diagnosis of placenta previa accreta according to RCOG criteria which are as follows) RCOG,2019):

2D greyscale signs: loss of myometrial interface or retroplacental clear space, reduced myometrial thickness, intra-placental blood flow and intra-placental lacunae.

2D color Doppler signs: intra-placental blood flow, the presence of altered blood flow in the retroplacental space and aberrant vessels crossing between placental surfaces.

All patients will be evaluated by ultrasonography examinations which will be performed at Ultrasound Special Care Unit Fetus, Ain Shams University Maternity Hospitals by ultrasound unit staff to confirm the gestational age, placental location. Lower placental edge thickness will be measured at the time of diagnosis using TVUS by the following technique. Visualization of lower placental edge will be done, while in the sagittal plane with the full length of the cervical canal and lower part of the uterus are in view. If the lower placental edge was not visualized, the transducer could be rotated 90° with the internal cervical os kept in view to detect the presence of placental tissue in the lower uterine cavity. Measurement of placental edge thickness of non-central placenta will be taken as the maximum measurement in the plane perpendicular to the long axis of the placenta, within 2cm of the lead point.

The thickness of the lower placental edge will be measured as the maximum thickness within a centimeter of the meeting point of the basal and chorionic plates. Thin placental edge will be considered when the thickness is <1cm. TVUS will be done at time of diagnosis to record measurement of lower placental edge thickness.

Follow-up of all cases and a scheduled elective cesarean section will be planned for all cases at completed 36 to 37 weeks of gestation following diagnosis of placental previa accreta by ultrasonography. Induction of fetal lung maturity will be carried out by giving 12 mg dexamethasone IM daily for two doses. If vaginal bleeding occurred prior to the scheduled cesarean section, patients will be admitted to the hospital and delivery will be decided in accordance with the clinical condition of the patient. Delivery will be performed at 36 completed weeks of gestation in cases of absent or mild vaginal bleeding. In cases of active bleeding that is clinically significant, or in those with massive APH, an emergency cesarean section will be done regardless of gestational age.

ELIGIBILITY:
Inclusion Criteria:

Single, viable gestations. Gestational age >28 weeks, < 36 weeks.

Confirmed diagnosis of placenta previa accreta when the placenta lies directly over the internal os based on ultrasound features among RCOG criteria as follows) RCOG,2019):

2D greyscale signs: loss of myometrial interface or retroplacental clear space, reduced myometrial thickness, intra-placental blood flow and intra-placental lacunae.

2D color Doppler signs: intra-placental blood flow, the presence of altered blood flow in the retroplacental space and aberrant vessels crossing between placental surfaces.

First time of diagnosis of placenta previa accreta is 28-30 weeks. Previous one or more cesarean sections.

Exclusion Criteria:

Maternal medical co-morbidities like diabetes and hypertension. Patients with bleeding disorders or anticoagulant therapy. Over distended uterus e.g.: multiple gestation, polyhydramnios, fetal macrosomia(>4.5kg).

Fetal anomalies or fetal growth restriction. Emergency cesarean section due to fetal distress. Rupture of membranes, intra-amniotic infection and fever during admission (>38 °C).

History of cervical cerclage or cervical cone biopsy.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: This study will be carried out on 50 women with a singleton pregnancy, between 28-36 weeks, with placenta previa accreta by suspected sonographic examination.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Lower placental edge thickness measurements by ultrasound in patients having placenta previa accreta. | Baseline
  Lower placental edge thickness measurements by ultrasound in patients having placenta previa accreta until delivery will occur.

SECONDARY OUTCOMES:
Type of cesarean delivery | Baseline
  elective versus emergency cesarean section <36 week of gestation due to massive hemorrhage
Gestational age at delivery. | Baseline
  Gestational age at time of delivery.
Antepartum bleeding, post-partum hemorrhage . | Baseline
  Antepartum bleeding, post-partum hemorrhage at the time of cesarean section.
Need for Cesarean hysterectomy | Baseline
  Need for Cesarean hysterectomy at time of delivery
Peripartum blood transfusion | Baseline
  Peripartum blood transfusion at time of delivery
Neonatal birth weight. | Baseline
  Neonatal birth weight at time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Fathi, MD, Study Director — World Health Organization
Locations (1):
- Ain Shams University Maternity Hospitals, Cairo, Egypt

REFERENCES:
- [Background] Syed W, Liaqat N, Naseeb G, Khattak SM. Relationship of placental edge thickness and cervical length to gestational age at delivery in patients with placenta previa. Pak J Med Sci. 2022 May-Jun;38(5):1349-1352. doi: 10.12669/pjms.38.5.5097. PMID 35799721
- [Background] Zaitoun MM, El Behery MM, Abd El Hameed AA, Soliman BS. Does cervical length and the lower placental edge thickness measurement correlates with clinical outcome in cases of complete placenta previa? Arch Gynecol Obstet. 2011 Oct;284(4):867-73. doi: 10.1007/s00404-010-1737-1. Epub 2010 Nov 27. PMID 21113721
- [Background] Jauniaux E, Alfirevic Z, Bhide AG, Belfort MA, Burton GJ, Collins SL, Dornan S, Jurkovic D, Kayem G, Kingdom J, Silver R, Sentilhes L; Royal College of Obstetricians and Gynaecologists. Placenta Praevia and Placenta Accreta: Diagnosis and Management: Green-top Guideline No. 27a. BJOG. 2019 Jan;126(1):e1-e48. doi: 10.1111/1471-0528.15306. Epub 2018 Sep 27. No abstract available. PMID 30260097